CLINICAL TRIAL: NCT03807713
Title: Clinical Study of Minimally Invasive Ponto Surgical Technique (MIPS) - Design Iteration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C69
Record Dates: First submitted 2019-01-08; First posted 2019-01-17 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2021-03

CONDITIONS: Bone Conduction Deafness; Unilateral Deafness; Middle Ear Deafness; Mixed Hearing Loss
MeSH Terms: conditions — Hearing Loss, Unilateral; Hearing Loss, Mixed Conductive-Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Minimally Invasive Ponto Surgery (Other): Surgical method for installation of a bone anchored hearing system for hearing rehabilitation
  Interventions: Device: Minimally Invasive Ponto Surgery

INTERVENTIONS:
Device: Minimally Invasive Ponto Surgery — Minimally Invasive Ponto surgery is used for hearing rehabilitation using Ponto Wide Implants in patients indicated and counselled for Bone Anchored Hearing Systems.

SUMMARY:
The objective of the study is to compare the outcomes after a surgical procedure with minimally invasive Ponto surgery (MIPS, test group) and tissue preservation surgery (control) for placing Oticon Medical Ponto implants and abutments.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Patient indicated for an ear level bone anchored sound processor.
* Healthy bone quality to allow for 4mm implant insertion.

Exclusion Criteria:

* Intraoperative switch to an alternative surgical technique
* Patients undergoing re-implantation (on the side being included in the study)
* Previous participation in the C47 study.
* Inability to participate in follow-up.
* Psychiatric disease in the medical history.
* Mental disability.
* Presumed doubt, for any reason, that the patient will be able to show up on all follow-ups.
* Diseases or treatments known to compromise the bone quality at the implant site, e.g. radiotherapy, osteoporosis, diabetes mellitus.
* Patients with natural skin height of >12mm (as there will be additional skin reduction needed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
Numbness (sensibility) around the implant | 6 months post surgery
  Total numbness around the implant will be assessed as a combination of gnostic and vital sensibility.

SECONDARY OUTCOMES:
Length of surgery | At surgery
  Compare the surgical time between test (this investigation) and control group (previous investigation, C47).
Unplanned visits | 36 months
  Investigate and compare the number of unplanned visits, including unplanned surgical procedures and other treatments for the test (this investigation) and control group (previous investigation, C47).
Adverse skin reactions | 36 months
  Investigate and compare the rate of adverse skin reactions using the Holgers Scale.
Adverse skin reactions | 36 months
  Investigate and compare the rate of adverse skin reactions using the IPS scale.
Pain perception by patient | 36 months
  Investigate and compare pain using a visual analogue scale 0-10
Implant survivability | 36 months
  Investigate and compare implant survivability in terms of reported implant loss.
Implant stability as measured with resonance frequency analysis, RFA. | 36 months
  Investigate and compare implant stability.
  Implant stability is monitored by measuring the implant stability quotient when following up on patients. Stability will be reported as implant stability quotient (ISQ).
Surgical wound healing time | 36 months
  Investigate and compare healing time after surgery.
  Follow-up visits after surgery will assess the healing of wound. This will be a yes/no assessment to be answered by the attending physician. The investigators will also evaluate skin reactions and record any medications that were given to aid in skin healing.
Wound dehiscence | 36 months
  Investigate wound dehiscence size after surgery.
Quality of Life Assessment | 36 months
  Investigate and compare subjective benefit as measured by SSQ questionnaire.
Quality of Life Assessment | 36 months
  Investigate and compare subjective benefit as measured by YORK questionnaire.
Quality of Life Assessment | 36 months
  Investigate and compare subjective benefit as measured by APHAB questionnaire.
Quality of Life Assessment | 36 months
  Investigate and compare subjective benefit as measured by GBI questionnaire.
Quality of Life Assessment | 36 months
  Investigate and compare subjective benefit as measured by GHSI questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Myrthe Hol, MD, PhD, Principal Investigator — Radboud UMC, Department of Otorhinolaryngology. The Netherlands
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No